CLINICAL TRIAL: NCT00664612
Title: Comparison of AirTraq Laryngoscope to Macintosh Laryngoscope for Intubation of Patients With Potential Cervical Spine Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: T. P. Turkstra, University of Western Ontario
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: R-07-337; 13481
Record Dates: First submitted 2008-04-18; First posted 2008-04-23 (Estimated); Last update posted 2008-10-16 (Estimated); Status verified 2008-10

CONDITIONS: Trauma
Keywords: Cervical Spine
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Air Traq then Macintosh
  Interventions: Device: AirTraq
- 2 (Experimental): Macintosh then AirTraq
  Interventions: Device: AirTraq

INTERVENTIONS:
Device: AirTraq — Laryngoscopy with AirTraq

SUMMARY:
Intubation is frequently required for trauma patients as part of the resuscitative effort. When the stability of the cervical spine is unknown, the potential for spinal cord damage during intubation is significant; the question of the safest intubating technique has not been resolved. Previous Studies have evaluated Macintosh Laryngoscopy, Bullard Laryngoscope, face mask ventilation, fibre-optic guided oral and nasal intubation, esophageal Combitube®, Laryngeal Mask Airway® (LMA), and Intubating Laryngeal Mask Airway® (ILMA) use with respect to cervical spine movement. Our previous study evaluated the Intubating Lighted Stylet (Lightwand®) and GlideScope® versus the Macintosh Laryngoscope.

Another method of securing endotracheal intubation, approved and in routine use, is the AirTraq® videolaryngoscope (ProMedic, Inc, Bonita Springs, FL, USA). The AirTraq videolaryngoscope is a videolaryngoscope with an external video display of the glottic opening and an endotracheal tube track to guide the ETT through the vocal cords (www.airtraq.com). When a clear view of the vocal cords is obtained, the endotracheal tube may be advanced into the trachea. This technique can be performed rapidly and safely and there is the perception that it involves less cervical spine movement than direct laryngoscopy.

We propose to study the AirTraq videolaryngoscope to determine if its use would result in reduced cervical spine movement during intubation.

DETAILED DESCRIPTION:
With the surgeon's consent, informed and written consent will be ob¬tained from patients who are undergoing elective surgery requiring general anesthesia with endotracheal intubation. Preoperative clinical assessment of the patients will include routine airway evaluation of dentition, mouth opening, tongue size, Mallampati score, and neck mobility, as well as height, weight, and age.

While awake, the patients will be placed on the operating room table with a rigid board under their head, neck, and torso in order to simulate the table on which patients involved in trauma are placed in the emergency room. In-line stabilization (ILS), as recommended by the ATLS guidelines, will be applied to maintain the patient's head in the neutral position and reduce neck movement dur¬ing laryngoscopy.

After standard pre-oxygenation, anesthesia will be induced in routine fashion with 2 3 mg/kg propofol and 2-5 mcg/kg fentanyl; rocuro¬nium 0.8 mg/kg will be administered to effect muscle paralysis. The patient will be then be ventilated with 100% O2 via bag/mask for 3 minutes. (Oxygenation with 100% O2 provides an oxygen reservoir for at least 5 minutes while laryngoscopy is completed.) This is the standard of care in anesthesia.

After the patient is anesthetized, a sealed envelope containing computer a generated random assignment will be opened. Laryngoscopy will then be performed two times, with the Macintosh laryngoscope and with the AirTraq videolaryngoscope, in random order as determined by the envelope. Between laryngoscopies, the patient will be ventilated with sevoflurane in 100% oxygen.

Male patients will be intubated with an 8.0 mm inner diameter endotracheal tube (ETT) and women with a 7.0 mm or 7.5 mm ETT at the discretion of the anesthesiologist.

For AirTraq videolaryngoscopy, the AirTraq will be inserted and a view of the vocal cords will be obtained. The ETT will be advanced through the track until the tip of the ETT is visible at the glottic opening and then removed with the AirTraq videolaryngoscope.

For direct Macintosh laryngoscopy, a size 3 laryngoscope blade will be recommended in all patients, but the anesthesiologist may choose another size if deemed necessary. With laryngoscopy, the glottis will be exposed to enable positioning of the endotracheal tube at the vocal cords.

During the second laryngoscopy in the above sequence, the trachea will be intubated. The study is then complete. The hard board will be removed and the surgery will proceed in the usual fashion.

The laryngoscopy and intubation will be recorded by a portable fluoroscopy unit for subsequent review by the radiologist to assess cervical spine movement.

Laryngoscopy time will be defined as the time from when the laryngoscope blade or AirTraq videolaryngoscope passes the teeth of the patient until the time the endotracheal tube is positioned at the opening of the larynx. If the intubation sequence is longer than 120 seconds, it will be deemed a failure and recorded as such.

The Cormack-Lehane score, representing the degree of glottic exposure, of the larynx will be recorded for all patients. Blood oxygen saturation, heart rate, and blood pressure will be recorded every minute during the study.

To minimize inter-operator variability, all bag-mask ventilation, laryngoscopy, and intubation will be completed by one person.

ELIGIBILITY:
Inclusion Criteria:

* Elective non-cardiac surgery patients requiring intubation for the surgery.
* (Cardiac surgery uses TEE; there would not be space for the fluoroscopy machine.)
* ASA 1-3
* Body Mass Index (BMI) < 35

Exclusion Criteria:

* patients with previous neck surgery or unstable C-spine
* patients with Reflux disease (GERD)
* patients who are or may be pregnant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-01; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
Cervical Spine Movement | Intubation

SECONDARY OUTCOMES:
Time to Intubation | Intubation

CONTACTS AND LOCATIONS:
Overall Officials: Timothy P Turkstra, MD, Principal Investigator — Western University, Canada
Locations (1):
- University of Western Ontario, London, Ontario, Canada